CLINICAL TRIAL: NCT06999824
Title: Revisiting the Concept of Nerve Sparing Radical Hysterectomy
Acronym: Neuro-Nerve
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#57/20
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancers
Keywords: cervical cancer; radical hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nerve sparing radical hysterectomy: Patients undergoing nerve sparing radical hysterectomy

SUMMARY:
Nerve-sparing radical hysterectomy aims to preserve the autonomic innervation of pelvic organs. In most studies, the preservation of the parasympathetic component of pelvic innervation is achieved by sparing the lymphovascular-neural tissue located at the base of the lateral paracervical tissue. This study explores an alternative surgical technique based on a different anatomical pathway of parasympathetic fibers, running more cranially and deeply within the pararectal space.

DETAILED DESCRIPTION:
The concept of preserving pelvic autonomic innervation during radical hysterectomy was first introduced by Yabuki, who emphasized the relevance of pelvic neuroanatomy in supporting nerve-sparing techniques. His work laid the foundation for later studies aiming to establish a reproducible surgical method for preserving both sympathetic and parasympathetic pathways. Anatomically, there is broad consensus regarding the course of the hypogastric (sympathetic) nerves and the strategies to preserve them during radical hysterectomy. However, there is no complete consensus regarding the preservation of parasympathetic fibers. Most current techniques derive from the approach described by Shingo Fujii in 2008, which involves the identification of the deep uterine veins within the lateral paracervical tissues to preserve the lymphovascular and parasympathetic fibers situated between the deep uterine vein and the pelvic wall.

However, in 2004, Raspagliesi et al. introduced a novel anatomical consideration, postulating the existence of two distinct groups of parasympathetic fibers-both originating from the sacral roots (S2-S4). The first group (named Group A) corresponds to the fibers preserved in the Fujii technique. The second group (named Group B) comprises three distinct fiber bundles running on a more cranial plane, within the pararectal space. The anatomical presence of these Group B fibers was initially reported by Baader and Herrmann in 2003; although without a precise description of their anatomical landmarks or functional significance. In the Raspagliesi et al. studises, both fiber groups were identified; however, Group A fibers were routinely resected to maintain the standard C2-type radical hysterectomy technique, which allowed for a shorter operative time. Conversely, Group B fibers were preserved without compromising bladder functional recovery. Current evidence suggests that postoperative bladder and rectal functional outcomes are comparable between the two approaches, indicating that preservation of Group A fibers may not be essential for maintaining pelvic autonomic function.

Most published studies based on the Fujii technique focus on preserving Group A fibers while overlooking the existence or relevance of Group B fibers, which often lie outside the standard surgical field and thus remain intact by default. This lack of anatomical and neurofunctional data on Group B has led some authors, including Muallem, to question their existence altogether.

Although intraoperative neurophysiological techniques have significantly evolved in recent decades, their application to pelvic autonomic nerve assessment remains limited due to the need for specialized protocols and a lack of standardized methodologies. Of note, no electrophysiology studies confirmed the value of preserving Group A fibers, thus highlighting the importance of further investigating the functional role of Group B fibers in maintaining pelvic autonomic function.

To address this gap, we designed a prospective study to test the hypothesis that the second group of parasympathetic fibers (Group B) does indeed exist and is functionally capable of autonomously innervating pelvic effector organs (bladder and rectum). Using intraoperative neurophysiological monitoring (IONM) and cystometry, we aim to assess the functional role of pelvic splanchnic nerves in autonomic control during nerve-sparing radical hysterectomy. Our findings may support the adoption of a safer and more effective nerve-sparing surgical technique by validating the role of these deeper parasympathetic fibers.

ELIGIBILITY:
Inclusion Criteria: (i) age ≥18 years; (ii) histologically confirmed cervical cancer; (iii) indication for type C1 (nerve-sparing) radical hysterectomy according to ESGO guidelines; and (iv) a minimum of 90 days of postoperative follow-up. Exclusion Criteria: (i) withdrawal of consent; (ii) prior abdominal and/or pelvic surgery; (iii) pre-existing urinary incontinence, detrusor overactivity, or detrusor underactivity; and (iv) pre-existing anorectal dysfunction Staging and architectural grade were defined according to the 2018 International Federation of Gynecology and Obstetrics (FIGO) recommendations, and histological subtypes were classified based on the World Health Organization (WHO) criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with cervical cancer
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Bladder dysfunction | 90 day after surgery
  Bladder dysfunction following radical hysterectomy is typically defined as any postoperative impairment in bladder storage or emptying function, which may include: Delayed or incomplete bladder emptying Increased post-void residual volume (PVR). Detrusor underactivity or acontractility Urinary retention requiring catheterization Loss of sensation of bladder fullness Urinary urgency, frequency, or incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Grazia Casadei, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano; Valentina Chiappa, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Will be share data only at the end of teh study